CLINICAL TRIAL: NCT02263482
Title: Inspiratory Muscle and Peripheral Muscle Combined Training Effects on the Respiratory and Functional Capacity and Quality of Life in Chronic Heart Failure
Brief Title: Inspiratory Muscle and Peripheral Muscle Training in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naomi Kondo Nakagawa (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Sponsor-Investigator, Naomi Kondo Nakagawa, Associate Professor of Medical School of Sao Paulo University, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 232/12; FAPESP 2013/13598-1 (Other Grant/Funding Number: Fundação de Amparo à Pesquisa do Estado de São Paulo)
Record Dates: First submitted 2014-09-29; First posted 2014-10-13 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Heart Failure
Keywords: muscle training; walking test; chronic heart failure; functional capacity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Other): patients awaiting for evaluation to cardiac rehabilitation or transplantation
  Interventions: Other: control
- moderate-intensity group (Experimental): Patients will be submitted to a 8-weeks training program, with inspiratory muscle trained at 30% of the maximal inspiratory pressure (30 minutes/session/7 days/week) and peripheral muscle trained with upper and lower exercises (50% of the 1-maximum repetition test).
  Interventions: Other: moderate-intensity group
- low-intensity group (Active Comparator): Patients will be submited to a 8 weeks training program, with inspiratory muscle trained at 15% of the maximal inspiratory pressure (30 minutes/session/7 days/week) and peripheral muscle trained with exercises of upper limbs and lower limbs (0,5 Kg each).
  Interventions: Other: low-intensity group

INTERVENTIONS:
Other: control — No intervention during the 8-weeks period of the study because of awaiting evaluation for cardiac rehabilitation or transplantation
  Arms: Control group
Other: moderate-intensity group — Patients will be submitted to a 8-weeks training program with inspiratory muscle trained at 30% of the maximal inspiratory pressure (30 minutes/session/7 days/week) + peripheral muscle trained with exercises of upper limbs and lower limbs (50% 1 RM, increased every 2-weeks).
  Arms: moderate-intensity group
Other: low-intensity group — Patients will be submited to a 8 weeks training program, with inspiratory muscle trained at 15% of the maximal inspiratory pressure (30 minutes/session/7 days/week) + peripheral muscle trained with exercises of upper limbs and lower limbs (0,5 kg each)
  Arms: low-intensity group

SUMMARY:
Heart failure is a clinical syndrome that is the common end of several cardiac diseases with symptoms such as muscle fatigue, dyspnea and reduction of quality of life. To improve respiratory and general functional capacity of these patients, there are strategies that can be used such as inspiratory muscle training and peripheral muscle training (dynamic resistance training).

DETAILED DESCRIPTION:
After agreement with the written informed consent, 35 subjects with severe heart failure were included in this study. They were randomized in three groups: controls, low-intensity and moderate-intensity group. All volunteers were assessed at Baseline and 8-weeks intervention. Cardiac events were registered following two years from baseline. The present study aimed to assess the effects of a combined program of inspiratory and peripheral muscle training on respiratory and general functional capacity and quality of life in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure (functional class from NYHA II and III),
* left ventricle ejection fraction bellow or equal 40%.

Exclusion Criteria:

* uncontrolled arrhythmia
* pulmonary edema or pulmonary congestion in the last 30 days
* peripheral oxygen saturation bellow 92% in resting condition
* respiratory infection in the previous 30 days to the enrollment into the study
* cognitive, neurological or orthopedic limitations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in respiratory muscle strength (in centimeters of water) | Before and after 8-weeks
  Inspiratory and expiratory muscle strength was assessed by using a pressure transducer (MVD-300 Microhard System, GlobalMed, Porto Alegre, Brazil).

SECONDARY OUTCOMES:
walking distance | Before and after 8-weeks
  To assess functional capacity using walking distance (6-min walk test accordingly to ATS and ERS guidelines)

OTHER OUTCOMES:
Change in pulmonary function | Before and after 8-weeks
  Pulmonary function will be assessed by spirometry.
Change in functional capacity | Before and after 8-weeks
  1RM
Inflammation in the upper airway by cytokines in blood | Before and after 8-weeks
  MMP2, myoglobin, p-selectin, MPO, NGAL, sVCAM, IL-2, IL-3, IL-4, IL-8,MIP1-alpha, 17, VEGF by Multiplex analysis. Inflammatory cells in nasal lavage will be also investigated.
Change in heart rate variability (HRV) | Before and after 8-weeks
  HRV is obtained from the spectral analysis of R-R intervals obtained from a heart rate monitor (Polar, S810, Kempele, Finland)
Prevalence of cardiac events and arrhythmia | Before and after 8-weeks
  by a 24-hours holter system for continuous recording of ambulatory electrocardiographic signs
Change in international Physical Activity Questionnaire (IPAQ) | Before and after 8-weeks
  Patients will be classified as sedentary, irregularly active, active or verry active according to Matsudo's classification (2001).
Change in quality of life using Minnesota Questionnaire | Before and after 8-weeks
  by Short Form-36 and by Minnesota Living with Heart Failure Questionnaire
  - Minnesota living with heart failure questionaire: contains 21 questions of physical, social, economic and emotional aspects. Each question ranges from zero to five points, with a total score of 105 points which is the maximum severity degree related to personal perception of quality of life.
Change in brain natriuretic peptide (BNP) analysis | Before and after 8-weeks
  A blood sample of 5 ml will be collected in a tube and BNP measured

CONTACTS AND LOCATIONS:
Overall Officials: Naomi K Nakagawa, PhD, Principal Investigator — USP
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil